CLINICAL TRIAL: NCT00160355
Title: Haploidentical Hematopoietic Stem Cell Transplantation for Pediatric Patients With Wiskott-Aldrich Syndrome: A Pilot Study
Brief Title: Haploidentical Hematopoietic Stem Cell Transplantation Patients With Wiskott-Aldrich Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WASHAP
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2009-02

CONDITIONS: Wiskott-Aldrich Syndrome
Keywords: Wiskott-Aldrich Syndrome; Immunodeficiency; Haploidentical transplantation
MeSH Terms: conditions — Wiskott-Aldrich Syndrome; Immunologic Deficiency Syndromes | interventions — Hematopoietic Stem Cell Transplantation; fludarabine; Melphalan; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Procedure: Hematopoietic stem cell transplantation; Device: Miltenyi CliniMACS selection system; Drug: Fludarabine, Melphalan, Thiotepa

INTERVENTIONS:
Procedure: Hematopoietic stem cell transplantation — To determine the safety in regards to engraftment and toxicity within 100 days of infusing a haploidentical T- and B-cell depleted hematopoietic stem cell graft into patients with Wiskott-Aldrich syndrome who have received a reduced intensity conditioning regimen.
  Other Names: Haploidentical stem cell transplant; Allogeneic stem cell transplant; Mismatched family member donor transplant; T and B cell depletion
Device: Miltenyi CliniMACS selection system — This system depletes the hematopoietic stem cell graft of T and B lymphocytes.
Drug: Fludarabine, Melphalan, Thiotepa — Participants will receive a reduced intensity conditioning regimen consisting of Fludarabine, Melphalan, Thiotepa, and OKT3 prior to receipt of the haploidentical stem cell graft. Rituximab will be given in an effort to prevent PTLPD. In addition to T-cell depletion of the donor product, cyclosporine will be given for GVHD prophylaxis.

SUMMARY:
Wiskott - Aldrich syndrome (WAS) is a rare disorder curable only through allogeneic hematopoietic stem cell transplantation. A mismatched family member is an option when no human leukocyte antigen (HLA-immune system type) matched related or matched unrelated donor is available.

This study will evaluate a novel therapeutic strategy for patients with WAS who undergo haploidentical transplantation using a parental donor. To reduce the risk of transplant-related toxicities, participants will receive a reduced intensity chemotherapy and antibody regimen (conditioning treatment). Participants will then receive an infusion of donor stem cells depleted of certain white blood cells called T- and B-lymphocytes. The stem cell depletion processing will be done through the use of the investigational CliniMACS device. A certain number of T-lymphocytes will be added back to the processed stem cell graft prior to infusion into the recipient.

The primary objective of this study is to determine the safety of haploidentical transplantation in WAS patients using this specified conditioning regimen and engineered graft. Safety will be defined in terms of engraftment (meaning how well the graft grows and functions after infusion) and regimen-related toxicity within the first 100 days after transplant.

DETAILED DESCRIPTION:
Secondary Objectives in this trial include the following:

* To estimate the survival of study recipients at one year after infusion of the T- and B-lymphocyte depleted stem cell graft.
* To assess if the study treatment enables the recipient to generate normal donor-derived B-cell numbers and endogenous IgM, IgG, and IgA production, resulting in a reduction/elimination of the need for intravenous immunoglobulin infusions.
* To determine if the study treatment results in the ability of the research participant to generate normal donor-derived T cell response and natural killer (NK) cell numbers and function.
* To describe the incidence of Epstein-Barr virus-lymphoproliferative disease (EBV-LPD) in these transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Genotypical diagnosis of Wiskott-Aldrich Syndrome.
* Less than 18 years of age at time of transplant.

Must meet two of the eight following clinical criteria:

* Eczema that is refractory to standard therapy.
* Thrombocytopenia as defined by a platelet count < 50,000/mm3.
* Significant risk for or presence of opportunistic infection.
* Autoimmune disease.
* Malignancy or pre-malignant condition.
* Family history as defined as a family member with WAS who died before 10 years of age.
* Does not have a suitable, available 6/6 HLA-matched sibling donor available for donation.
* Does not have a suitable, available 10/10 HLA-allele matched unrelated donor identified through the National Marrow Donor Program (NMDP).

Exclusion Criteria:

If any of the following clinical indicators are met within 45 days prior to transplant, the research participant will not be eligible for the study:

* Symptomatic cardiac disease or evidence of significant cardiac dysfunction by echocardiogram (shortening fraction < 30%).
* Creatinine clearance or Tc 99 less than or equal 40ml/min/1.73 m2.
* SGPT greater than or equal 500 U/L.
* Karnofsky or Lansky Performance Score of < 50.
* Pulmonary function tests: FVC < 50% of predicted value if age appropriate to perform the testing adequately or an O2 saturation less than or equal to 92% on room air at rest.

Max Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2005-05; Primary Completion 2008-07 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To determine safety in regards to engraftment and toxicity within 100 days post-haploidentical T- and B-cell depleted hematopoietic stem cell transplantation for patients with Wiskott-Aldrich syndrome who received a reduced intensity conditioning | March 2010

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Kasow, DO, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org